CLINICAL TRIAL: NCT06215274
Title: The Impact of Cognitive Leisure Activity Levels on Cognitive Function in the Preclinical Stage of Alzheimer's Disease and the Study of Its Neural Circuitry Regulation Mechanisms
Brief Title: Cognitive Leisure and Preclinical Alzheimer's Disease: Exploring Neural Mechanisms
Status: Recruiting | Type: Observational
Sponsor: Yuanjiao Yan (Other)
Responsible Party: Sponsor-Investigator, Yuanjiao Yan, Principal Investigator, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Other Study IDs: K2023-12-004
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Dysfunction
Keywords: Alzheimer's Disease; Cognitive Leisure activity; MRI
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People in the stage of preclinical Alzheimer's disease: Observe the cognitive leisure activity levels, cognitive function, and MRI characteristics in patients in the preclinical stage of Alzheimer's Disease
  Interventions: Other: Relationship of the cognitive leisure activity levels, cognitive function, and MRI characteristics.

INTERVENTIONS:
Other: Relationship of the cognitive leisure activity levels, cognitive function, and MRI characteristics. — The cognitive leisure activity levels, cognitive function, and MRI characteristics in people in the preclinical stage of Alzheimer's Disease (AD).

SUMMARY:
The goal of this clinical trial is aims to:

1. Translate and culturally adapt the Cognitive Leisure Activity Scale (CLAS) into Chinese and Conduct reliability and validity tests for the Chinese version of CLAS.
2. Investigate the correlation between cognitive leisure activity levels and cognitive function in the preclinical stage of Alzheimer's Disease (AD).
3. Clarify the regulatory mechanisms of cognitive leisure activity levels on the neural circuits of patients in the preclinical stage of AD.

DETAILED DESCRIPTION:
Alzheimer's disease (AD), also known as senile dementia, is the most common neurodegenerative disorder characterized by progressive decline in cognitive function and behavioral impairment. It is estimated that there are approximately 9.83 million AD patients in China, with an average annual treatment cost of about $19,144 per person, accounting for 1.47% of the national gross domestic product, surpassing the global average. This not only severely affects the quality of life for elderly patients but also imposes a heavy economic and caregiving burden on families and society.

Due to the limitations of AD treatment and the irreversibility of its progression, early detection and intervention have become the focus of AD prevention and control efforts. Increasingly, scholars propose shifting the diagnosis and intervention of AD to the preclinical stage, particularly the mild cognitive impairment (MCI) phase and even earlier stages characterized by subjective cognitive decline (SCD). Cognitive leisure activity, as one of the potentially modifiable factors in the preclinical stage of AD, understanding its impact on cognitive function and the neural circuitry regulation mechanisms in this stage is of significant importance. This knowledge can contribute to the development of early targeted intervention measures, preventing or delaying the onset and progression of AD, and promoting healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Mild Cognitive Impairment (MCI) and Subjective Cognitive Decline (SCD)
* Age ≥ 60 years
* Capable of normal communication in Mandarin，possesses a certain level of comprehension and judgment.

Exclusion Criteria:

* Individuals with severe hearing or language impairments, or with severe physical illnesses that are unable to cooperate with the survey
* Individuals with pacemakers, metallic implants, cochlear implants, claustrophobia, and other contraindications for MRI examination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Older adults in the stage of preclinical AD
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive leisure activity levels | Baseline
  The Chinese version of Cognitive & leisure activity scale will be used. Utilizing the Likert 5-point scale with 16 items, total score ranges from 0 to 80 points，higher scores signify increased cognitive leisure activity levels. An abnormal level is determined if the score is below 25 points.

SECONDARY OUTCOMES:
Memory | Baseline
  The Chinese version of Auditory Verbal Learning Test will be used. This includes immediate memory, short-term memory, long-term memory, and recognition memory. A higher score indicates better memory performance.
Verbal fluency | Baseline
  The Chinese version of Verbal Fluency Test will be used. A higher score indicates better verbal language performance.
Executive function | Baseline
  The Chinese version of Shape Trail Test will be used. The shorter the usage time indicates better executive functioning.
Visuospatial skills | Baseline
  The Chinese version of Rey-Osterrieth Complex Figure Test will be used. A higher score indicates better visual-spatial structural abilities.
Naming difficulty | Baseline
  The Chinese version of Boston Naming Test will be used. The total scores range from 0 to 30, a higher score indicates better language functioning.
Amplitude of Low-Frequency Fluctuations | Baseline
  The rest-state functional MRI of Amplitude of Low-Frequency Fluctuations analysis will be performed to investigate the variations in MRI features across different cognitive leisure activities and levels of cognitive functioning.
Regional Homogeneity | Baseline
  The rest-state functional MRI of Regional Homogeneity analysis will be performed to investigate the variations in MRI features across different cognitive leisure activities and levels of cognitive functioning.
Functional Connectivity | Baseline
  The rest-state functional MRI of Functional Connectivity analysis will be performed to investigate the variations in MRI features across different cognitive leisure activities and levels of cognitive functioning.
General cognitive function | Baseline
  The Chinese version of Montreal Cognitive Assessment will be used.The scale has a total score of 30 points, encompassing eight assessment sections: visual-spatial and executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. It involves multiple cognitive domains. A higher score indicates better cognitive functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjiao Yan, PHD, Study Director — Fujian Provincial Hospital\Shengli clinical medical college of Fujian Medical university
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Research data and research-related materials will be available in a repository or online. After completion of the study, relevant data will be provided in the form of a URL or DOI.
Supporting Information: SAP, Analytic Code
Time Frame: After completion of the study, relevant data will be provided in the form of a URL or DOI.
Access Criteria: Researchers whose proposed use of the data has been approved